CLINICAL TRIAL: NCT00074646
Title: Phase I Trial of CC-8490 for the Treatment of Subjects With Recurrent/Refractory High-Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Organization: Celgene (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CC-8490-GLIO-001
Record Dates: First submitted 2003-12-17; First posted 2003-12-19 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2007-01

CONDITIONS: Glioblastoma; Malignant Gliomas
Keywords: CC-8490; CC8490; Glio; Glioblastoma; Malignant Gliomas
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — CC-8490

INTERVENTIONS:
Drug: CC-8490

SUMMARY:
Phase I trial of CC-8490 for the treatment of subjects with recurrent/refractory high-grade gliomas

ELIGIBILITY:
Inclusion Criteria:

* Patients with glioblastoma multiforme (GBM), gliosarcoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), malignant glioma/astrocytoma NOS (not otherwise specified). Also included will be radiographically diagnosed infiltrating brain stem gliomas not amenable to biopsy. Other CNS tumor histologies will not be eligible for this trial.
* Patients must have shown either evidence for tumor recurrence or progression by CT or (preferably) MRI scan performed within 21 days prior to registration or had biopsy proven recurrent glioma within the last 12 weeks prior to enrollment (in order to allow the enrollment of patients with recurrent gliomas who have undergone a complete radiographic resection and now have no radiographic evaluable disease)
* Patients having undergone recent resection of a recurrent or progressive tumor will be eligible two weeks after surgery.
* Patient must have failed prior radiation therapy and must have an interval of greater than or equal to 2 weeks from the completion of radiation therapy to study entry.
* All patients must sign an informed consent, or if cognitively impaired, their assigned DPA, indicating that they are aware of the investigational nature of this study.
* Patients must be > 18 years old, and must have a life expectancy > 8 weeks.
* Patients must have a Karnofsky performance status of > 60.
* Additionally, patients must be at least 6 weeks from nitrosoureas, 4 weeks from temozolomide or carboplatin, 3 weeks from procarbazine, and 2 weeks from last vincristine administration. Patients must be at least 4 weeks from other cytotoxic therapies not listed above and 2 weeks for non-cytotoxic agents (e.g., interferon, tamoxifen).
* Patients must have adequate bone marrow function (granulocyte count >= 1500/mm3, platelet count of > 100,000/mm3, and hemoglobin > 8 gm%), adequate liver function (total bilirubin <= 1.5 mg/dL, AST/ALT <= 2 x ULN), and adequate renal function (creatinine <= 1.5 mg/dL or creatinine clearance > 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion. Eligibility level for platelets may not be reached by transfusion.
* Patients must either not be receiving steroids, or be on a stable dose of steroids for at least five days prior to registration.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) are ineligible, unless they are in complete remission and off all therapy for that disease for a minimum of 3 years.
* Patients must not be pregnant or nursing, and all patients (both men and women) must be willing to practice birth control during and for 2 months after treatment with CC-8490. Women of childbearing potential (WCBP) who are sexually active must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).
* Patients must be able to swallow capsules whole.

Exclusion Criteria:

* Patients who, in the view of the treating physician, have significant active cardiac, hepatic, renal, or psychiatric diseases that would significantly increase the risk of using CC-8490 are ineligible.
* Concurrent use of other standard chemotherapeutics or investigative agents.
* Pregnant or lactating females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study, obscures the evaluation of toxicity or alters drug metabolism.
* Use of other experimental study drug within 28 days of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-12; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Locations (1):
- Neuro Oncology BranchNational Cancer Institute, Bethesda, Maryland, United States